CLINICAL TRIAL: NCT00970619
Title: Ultrasound Accelerated Catheter-directed Thrombolysis for Primary Iliofemoral Deep Vein Thrombosis (IFDVT) Compared to Non-invasive Conventional Anticoagulant Therapy Alone: a Dutch Randomized Controlled Multicenter Clinical Trial
Brief Title: DUTCH CAVA-trial: CAtheter Versus Anticoagulation Alone for Acute Primary (Ilio)Femoral DVT.
Acronym: NL28394
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MEC 09-2-093
Record Dates: First submitted 2009-09-01; First posted 2009-09-02 (Estimated); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Acute Thrombosis of Deep Veins of Proximal Lower Extremity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional anticoagulation therapy (No Intervention): Conservative treatment consists of an initial treatment with therapeutic doses of low molecular weight heparin (LMWH) in combination with vitamin K-antagonists, followed by treatment with vitamin K-antagonist alone (after completing LMWH treatment of at least 5-7 days and after an international normalized ratio (INR) above 2 has been reached on two consecutive measurements). Or alternatively the new direct activated factor X inhibitors can be used as anticoagulation therapy. Anticoagulant treatment will be installed according to national and international guidelines (ACCP 2008 [23], CBO 2008 [24]) tailored based on the character of the event (6 months of therapy for idiopathic DVT and 3 months for provoked DVT).
- Ekos Endowave system thrombolysis (Experimental): Catheter directed thrombolysis will be performed with an Ekos Endowave ® system (EKOS Corporation, Bothell, WA). The system uses a standard guide wire to position the Intelligent Drug Delivery Catheter across the length of the target clot. The guide wire is introduced through the popliteal vein. Along the guide wire the catheter is positioned. The location of the dispersion catheter is controlled and if necessary adjusted by X-ray. The guide wire is then pulled out and replaced with the Microsonic core (a miniscule high frequency (2MHz) ultrasound transducer). The system automatically monitors and controls the microsonic energy delivery. This system does not fragment the thrombus but only gives a structural change by which a better penetration of the thrombolytic agent is achieved.
  Interventions: Device: Ekos endowave system thrombolysis

INTERVENTIONS:
Device: Ekos endowave system thrombolysis — Catheter directed thrombolysis will be performed with an Ekos Endowave ® system (EKOS Corporation, Bothell, WA). The system uses a standard guide wire to position the Intelligent Drug Delivery Catheter across the length of the target clot. The guide wire is introduced through the popliteal vein. Along the guide wire the catheter is positioned. The location of the dispersion catheter is controlled and if necessary adjusted by X-ray. The guide wire is then pulled out and replaced with the Microsonic core (a miniscule high frequency (2MHz) ultrasound transducer). The system automatically monitors and controls the microsonic energy delivery. This system does not fragment the thrombus but only gives a structural change by which a better penetration of the thrombolytic agent is achieved.
  Other Names: Ekos endowave ® system
  Arms: Ekos Endowave system thrombolysis

SUMMARY:
Rationale: Iliofemoral deep venous thrombosis (IFDVT) is associated with significant post thrombotic morbidity. The presence of both obstruction and reflux significantly increases the chances for development of post-thrombotic syndrome (PTS). Early thrombolysis may reduce the incidence of PTS as compared to treatment with conventional anticoagulant medication alone. Improvement of the health related quality of life (HRQOL) has been reported after surgical clot removal. The investigators hypothesize that such improvements could also be reached after catheter-directed thrombolysis (CDT).

Objective: To assess whether CDT for the treatment of IFDVT can safely and effectively reduce post-thrombotic morbidity after one year. The secondary objective is to study whether CDT intervention has a positive effect on the HRQOL of patients with IFDVT and to assess late PTS.

Study design: Prospective, multicenter, single-blind, allocation concealed, randomized controlled trial Study population: All consecutive patients with IFDVT presenting at the emergency or outpatient departments of the participating centers. The thrombus should not be older than 14 days at randomization.

Intervention: After randomization patients will be allocated to either conservative anticoagulant treatment or to CDT combined with conservative anticoagulant treatment.

Main study parameters/endpoints: The primary efficacy outcome is the proportion of PTS at one year; a decline in PTS incidence from 25% to 8% is anticipated. The secondary outcome is the Health related Quality of life. The principal safety outcome is major bleeding during anticoagulant therapy. Bleeding as well as events of recurrent thrombosis will be monitored. Measurements of markers of coagulation and inflammation will be performed during follow-up. After CDT the patency of the venous system in the affected lower limb will be assessed as well as the percentage of clot lysis. The development of late PTS during follow-up will also be monitored.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: For patients who are randomized to CDT a hospital stay for 24-96 hours is mandatory. All patients will undergo additional imaging by magnetic resonance venography and air phletysmography (if available) at baseline and after 12 months; blood will be taken at these visits. Clinical follow-up visits will be matching usual care at 3, 6, 12 months. Health-related quality of life (HRQOL) questionnaires will be filled out by all patients at baseline, 3, 6 and 12 months after the event; and once a year during the entire study duration. Further treatment will be in accordance with current guidelines for antithrombotic treatment. There may be an enhanced risk of bleeding in the thrombolysis group. The expected benefit is reduction of PTS from 25% to 8%, together with an improved quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Objectively documented IFDVT
* Acute stage IFDVT, complaints less than 14 days
* Life expectancy longer than 6 months
* First thrombus in the affected limb

Exclusion Criteria:

* History of GI bleeding within 1 year
* History of cardiovascular accident /central nervous system disease within 1 year
* Severe hypertension (>180/100 mmHg)
* Active malignancy
* Major surgery within 6 weeks
* Previous thrombosis of the affected limb (secondary thrombosis)
* Varicosities/venous insufficiency Clinical, Etiologic, Anatomic, and Pathophysiologic (CEAP) classification C3 or higher
* Pregnancy
* Immobility (wheelchair dependent)
* Alanine aminotransferase (ALAT) > 3 times normal range
* estimated Glomerular Filtration Rate (eGFR) < 30 mL/min

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2010-05 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Post thrombotic syndrome (percentage of patients with PTS) one year following the acute thrombotic event. | one year

SECONDARY OUTCOMES:
The Health Related Quality of Life (HRQOL) | 5 years
PTS during follow-up | 5 years
Recurrent venous thrombo-embolisms (VTE): DVT/Pulmonary Embolism during follow-up | 5 years
Clot lysis, patency and valve function | 5 years
Measurements of markers of coagulation and inflammation | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Hugo ten Cate, MD, PhD, Principal Investigator — Maastricht University Medical Centre
Locations (16):
- Netherlands (16):
  - Maastricht University Medical Centre, Maastricht, Limburg
  - Academisch Medisch Centrum, Amsterdam
  - VuMC, Amsterdam
  - Nij Smellinghe, Drachten
  - Catharina Ziekenhuis Eindhoven, Eindhoven
  - MMC Eindhoven, Eindhoven
  - St Anna Ziekenhuis, Geldrop
  - Atrium MC Heerlen, Heerlen
  - Elkerliek Ziekenhuis, Helmond
  - St Antonius, Nieuwegein
  - Laurentius Roermond, Roermond
  - Maasstad ziekenhuis, Rotterdam
  - Haga Ziekenhuis, The Hague
  - VieCuri, Venlo
  - Sint Jans Gasthuis, Weert
  - Isala klinieken, Zwolle

REFERENCES:
- [Derived] Flumignan RL, Nakano LC, Flumignan CD, Baptista-Silva JC. Angioplasty or stenting for deep venous thrombosis. Cochrane Database Syst Rev. 2025 Feb 19;2(2):CD011468. doi: 10.1002/14651858.CD011468.pub2. PMID 39968829
- [Derived] Iding AFJ, Alkarithi G, Cate HT, Ariens RAS, Ten Cate-Hoek AJ. Fibrinogen levels and clot properties identify patients who benefit from catheter-directed thrombolysis after DVT. Blood Adv. 2024 Jun 11;8(11):2924-2932. doi: 10.1182/bloodadvances.2023012493. PMID 38547453
- [Derived] Arnoldussen CWKP, Notten P, Brans R, Vroegindeweij D, Tick LW, van de Poel MHW, Wikkeling ORM, Vleming LJ, Koster A, Jie KG, Jacobs EMG, Planken N, Wittens CHA, Ten Cate H, Wildberger JE, Ten Cate-Hoek AJ. Clinical impact of assessing thrombus age using magnetic resonance venography prior to catheter-directed thrombolysis. Eur Radiol. 2022 Jul;32(7):4555-4564. doi: 10.1007/s00330-022-08599-5. Epub 2022 Mar 28. PMID 35347362
- [Derived] Notten P, de Smet AAEA, Tick LW, van de Poel MHW, Wikkeling ORM, Vleming LJ, Koster A, Jie KG, Jacobs EMG, Ebben HP, Coppens M, Ten Cate H, Wittens CHA, Ten Cate-Hoek AJ. CAVA (Ultrasound-Accelerated Catheter-Directed Thrombolysis on Preventing Post-Thrombotic Syndrome) Trial: Long-Term Follow-Up Results. J Am Heart Assoc. 2021 Jun;10(11):e018973. doi: 10.1161/JAHA.120.018973. Epub 2021 May 25. PMID 34032127
- [Derived] Notten P, Arnoldussen CWKP, Brans R, de Smet AAEA, Tick LW, van de Poel MHW, Wikkeling ORM, Vleming LJ, Koster A, Jie KG, Jacobs EMG, Ebben HP, Planken N, Ten Cate H, Wittens CHA, Ten Cate-Hoek AJ. Association of Successful Ultrasound-Accelerated Catheter-Directed Thrombolysis with Postthrombotic Syndrome: A Post Hoc Analysis of the CAVA Trial. Thromb Haemost. 2020 Aug;120(8):1188-1199. doi: 10.1055/s-0040-1713171. Epub 2020 Jun 30. PMID 32604427
- [Derived] Notten P, Ten Cate-Hoek AJ, Arnoldussen CWKP, Strijkers RHW, de Smet AAEA, Tick LW, van de Poel MHW, Wikkeling ORM, Vleming LJ, Koster A, Jie KG, Jacobs EMG, Ebben HP, Coppens M, Toonder I, Ten Cate H, Wittens CHA. Ultrasound-accelerated catheter-directed thrombolysis versus anticoagulation for the prevention of post-thrombotic syndrome (CAVA): a single-blind, multicentre, randomised trial. Lancet Haematol. 2020 Jan;7(1):e40-e49. doi: 10.1016/S2352-3026(19)30209-1. Epub 2019 Nov 27. PMID 31786086